CLINICAL TRIAL: NCT01939145
Title: A Prospective Randomized Trial Comparing Outcomes for Prontosan Versus Normal Saline for Negative Pressure Wound Therapy With Instillation
Brief Title: Comparing Outcomes for Prontosan Versus Normal Saline for Negative Pressure Wound Therapy With Instillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Paul J. Kim, DPM, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06142013
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Wound Infection
Keywords: hospital admission
MeSH Terms: conditions — Wound Infection | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Active Comparator): The use of Normal Saline as the solution for Negative Pressure Wound Therapy with instillation.
  Interventions: Drug: Normal saline
- Prontosan (Active Comparator): The use of Prontosan as the solution in Negative Pressure Wound Therapy with Instillation.
  Interventions: Device: Prontosan

INTERVENTIONS:
Drug: Normal saline — Normal saline (0.9% NaCl) is an isotonic solution that is widely used for intravenous application but is also used as our SOC for wound irrigation. This solution has high tolerability. Normal saline has been used as the instillation solution for NPWTi. The dwell setting for this solution is 20 minutes. The volume of solution to be used is dependent on the size of the wound hence varies
  Other Names: 0.9% Saline
  Arms: Normal Saline
Device: Prontosan — Prontosan (B Braun, Bethlehem, PA) is 0.1% polyhexanide, 0.1% betaine, sodium hydroxide, and purified water. The polyhexanide is an antiseptic and betaine is a surfactant. This solution is an FDA approved device indicated for topical irrigation. This solution has high tolerability with robust antimicrobial activity. Polyhexanide has been utilized as the instillation solution for NPWTi with positive clinical results. Prontosan is currently being used as the instillation solution for NPWTi in this facility as the SOC. The dwell setting for this solution is 20 minutes. The volume of solution to be used is dependent on the size of the wound hence varies.
  Other Names: Prontosan Wound Irrigation Solution
  Arms: Prontosan

SUMMARY:
This is a prospective, randomized trial comparing the outcomes for Prontosan versus normal saline as the solution for negative pressure wound therapy with instillation (NWPTi). Negative pressure wound therapy (NPWT) is a well established method of treatment for acute and chronic wounds. The combination of negative pressure with instillation of a solution is a relatively novel concept that has gained popularity and is currently used nationally and internationally. NPWTi is the standard of care for our division. Despite the growing use, there is limited information regarding the selection of the ideal instillation solution. This is a single site, investigator initiated, NPWTi study comparing the use of Prontosan with normal saline for the adjunctive treatment of the acutely infected wound that requires hospital admission. A total of 100 subjects will be included with 50 subjects in each treatment arm. The outcomes that will be measured are 1) number of operations, 2) length of hospital stay, 3) % of wounds closed prior to discharge, 4) time to closure prior to discharge, 5)% remained closed at 30 day follow-up, and 6) reduction of qualitative bacterial cultures. The results from this study will better characterize the most appropriate use of NPWTi.

DETAILED DESCRIPTION:
Overview This is a prospective, randomized, comparative trial examining 2 different instillation solutions for NPWTi. All wound types that meet the eligibility criteria will be enrolled into the study. After enrollment, subjects will be randomized into either the Prontosan NPWTi group (n=50) or the normal saline NPWTi group (n=50). Data will be collected from inpatient hospital records.

Outline of Study Procedures

1. Patients meeting the eligibility criteria requiring hospital admission for an infected wound will be identified. Demographic information will be obtained.
2. Informed consent will be obtained.
3. Subjects will be taken to the operating room for wound debridement within 72 hours of admission per standard of care (SOC). Further, antibiotic therapy and medical management will be performed per SOC.
4. Randomization into the Prontosan or normal saline instillation group will be conducted after the informed consent has been signed, but before the first operation.
5. For the first operating room visit the following will be conducted:

   1. Pre- and post debridement qualitative cultures
   2. Debridement performed in SOC fashion
   3. Post debridement measurements
   4. Application of NPWTi
6. For subsequent operating room visits the following will be conducted:

   a. Pre- and post debridement qualitative cultures b. Debridement performed in SOC fashion c. Post debridement measurements d. Application of NPWTi or closure i. The decision to close the wound will be determined by the clinician per SOC.

   ii. The technique utilized for closure will be determined by the clinician per SOC.
7. Subjects will discharged from the hospital

   a. Criteria for discharge will be per the judgment of the investigator per SOC
8. After hospital discharge, the subject will be followed in the outpatient wound clinic per SOC. Information from the one month follow-up period will be collected. Subjects will be exited from the study at that point.

Subject Recruitment No active recruitment strategy will be employed. Patients who meet the eligibility criteria will be approached to participate into the study.

Participation Completion and Discontinuation:

Subjects may elect to discontinue participation at any time for any reason. Investigators may elect to remove the subject from participating at any time for any reason.

Surgical Technique:

Surgical debridement will be performed in SOC manner and is at the discretion of the investigator.

Postoperative Care:

Will be conducted in customary SOC fashion and is at the discretion of the investigator. The 30 day follow-up visit is part of SOC

Application of Devices/Dressing:

The device that will be utilized is the V.A.C. Ulta with Veraflo Technology (Kinetic Concepts Inc., San Antonio, TX). This is an FDA approved device that is indicated for wound care. The investigators currently use this device as the SOC for the inpatient management of the acutely infected wound. The device consists of a foam sponge applied to the wound surface with an adhesive drape that keeps it in place. This device applies subatmospheric pressure at -125mmHg to the wound surface. The instillation component includes the delivery of a topical solution at prescribed fashion to the wound surface. This solution is dwelled (no negative pressure during this interval) in the sponge for a specific duration and then is evacuated.

Negative Pressure Wound Therapy:

The setting for negative pressure will be -125mmHg, continuous setting, and moderate intensity. The application of the foam and drape will be conducted in the customary fashion. The negative pressure duration will be 2 hours.

Prontosan:

Prontosan (B Braun, Bethlehem, PA) is 0.1% polyhexanide, 0.1% betaine, sodium hydroxide, and purified water. The polyhexanide is an antiseptic and betaine is a surfactant. This solution is an FDA approved device indicated for topical irrigation. This solution has high tolerability with robust antimicrobial activity. Polyhexanide has been utilized as the instillation solution for NPWTi with positive clinical results. Prontosan is currently being used as the instillation solution for NPWTi in this facility as the SOC. The dwell setting for this solution is 20 minutes. The volume of solution to be used is dependent on the size of the wound hence varies.

Normal Saline:

Normal saline (0.9% NaCl) is an isotonic solution that is widely used for intravenous application but is also used as our SOC for wound irrigation. This solution has high tolerability. Normal saline has been used as the instillation solution for NPWTi. The dwell setting for this solution is 20 minutes. The volume of solution to be used is dependent on the size of the wound hence varies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than 18 years of age
* Admission to the hospital for an infected wound
* Diabetic, ischemic, neuropathic, venous, surgical wounds, any anatomical location
* Subjects requiring serial (more than 1) operative debridement

Exclusion Criteria:

* Pregnancy
* Patients with exposed bowel, brain matter, spinal cord
* Patients with exposed peripheral bypass grafts
* Known allergy or sensitivity to Prontosan or components of NPWT
* Known allergy or sensitivity to adhesives
* Uncontrolled bleeding disorders/coagulopathy
* Wounds that tunnel to unexposed areas
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kim, DPM, Study Director — MedStar Georgetown University Hospital; Christopher Attinger, MD, Principal Investigator — MedStar Georgetown University Hospital; John Steinberg, DPM, Principal Investigator — MedStar Georgetown University Hospital; Karen Evans, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital Center for Wound Healing, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data collected has not been approved for use beyond the scope of this trial and will not be made available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline | Prontosan
Started | 49 | 51
Completed | 47 | 44
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Prontosan | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.64 (15.4) | 55.94 (13.9) | 58.37 (14.09)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 8 | 29
  Male | 28 | 43 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  African America | 21 | 21 | 42
  Caucasian | 22 | 23 | 45
  Asian | 1 | 5 | 6
  Hispanic | 2 | 1 | 3
  Other | 1 | 0 | 1
  Missing/declined | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Operating Room Visits
Description: Compare the number of operative room visits between Prontosan NPWTi and normal saline NPWTi.
Time Frame: Patients will be followed during their hospital stay which is an average of approximately 2 weeks.
Measure: Mean (Standard Deviation); unit: Operative Room Visits
Arm/Group | Normal Saline | Prontosan
Number analyzed (Participants) | 49 | 51
Operative Room Visits | 2.5 (0.9) | 2.8 (0.9)

2. Secondary Outcome: Hospital Admission Length of Stay
Description: Compare the hospital admission length of stay between Prontosan NPWTi and normal saline NPWTi.
Time Frame: Patients will be followed during their hospital stay which is an average of approximately 2 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Normal Saline | Prontosan
Number analyzed (Participants) | 49 | 51
days | 13.6 (11.7) | 14.5 (9)

3. Other Pre Specified Outcome: Time to Closure
Description: Compare the percent of wounds closed and the time to closure during the hospital admission and up to one year after discharge between Prontosan NPWTi and normal saline NPWTi.
Time Frame: Patients will be followed during their hospital stay which is an average of approximately 2 weeks.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Wound Recidivism
Description: Compare the percent of wounds that remained closed 30 days and up to one year after discharge between Prontosan NPWTi and normal saline NPWTi.
Time Frame: 30 days post discharge from hospital
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Bacterial Culture Results
Description: Compare the qualitative bacterial culture results between Prontosan NPWTi and normal saline NPWTi.
Time Frame: Patients will be followed during their hospital stay which is an average of approximately 2 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Normal Saline | Prontosan
Serious Adverse Events (participants affected / at risk) | 2/49 | 3/51
Other Adverse Events (participants affected / at risk) | 14/49 | 23/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=49) | Prontosan (N=51)
Amputation (Surgical and medical procedures) | 1 (1) | 3 (3)
Death (Cardiac disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=49) | Prontosan (N=51)
Infection (Infections and infestations) | 8 (9) | 9 (10)
Wound dehiscence (Surgical and medical procedures) | 6 (7) | 14 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes